CLINICAL TRIAL: NCT07176364
Title: Body Temperature Monitoring and Factors Affecting Body Temperature in Preterm Neonates Receiving Respiratory Support: Creating a Data Model
Brief Title: Body Temperature in Preterm Neonates: Creating a Data Model
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assoc. Prof., Acibadem University
Other Study IDs: ATADEK-2025/05
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Temperature; Preterm
Keywords: PRETERM; TEMPERATURE; INFANT; DECISION TREE; VENTILATION
MeSH Terms: conditions — Premature Birth; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infant: Preterm infants born before 38 weeks of gestation who were immediately admitted to the neonatal intensive care unit after birth and received respiratory support.

SUMMARY:
The aim of this study is to examine the relationship between the characteristics, medical history, interventions performed within the first six hours, and follow-up findings of preterm newborns receiving respiratory support and their body temperature. In this context, the aim was to establish a basic data model that would contribute to the optimization of practices aimed at maintaining thermoregulation in newborns receiving respiratory support.

H1: The characteristics, medical history, and variables related to the interventions performed in preterm newborns receiving respiratory support have a statistically significant relationship with body temperature.

H2: The developed data model can accurately and meaningfully predict the relationship between the characteristics, medical history, and interventions affecting body temperature in preterm newborns receiving respiratory support.

DETAILED DESCRIPTION:
Because the systems of preterm infants are not functionally mature, deficiencies are seen in critical physiological processes such as respiration and thermoregulation. Since respiratory functions are not fully developed, increased respiratory effort can increase energy expenditure and metabolic load, making it difficult to regulate body temperature and facilitate postnatal adaptation.

Increased respiratory effort can create a metabolic load that may increase the risk of hypothermia in preterm infants. In preterm infants experiencing respiratory distress, energy consumption increases, while the energy reserves necessary to maintain body temperature may be depleted more rapidly. As a result, thermoregulation may not be maintained, and the risk of hypothermia may increase. Furthermore, factors that increase respiratory effort may elevate oxygen demand, leading to changes in blood circulation and disruption of thermoregulatory mechanisms.

Maintaining normothermia in newborns is critically important and is known to have a direct impact on survival. The World Health Organization recognizes maintaining normothermia as a fundamental and critical component of newborn care.

Studies have shown that respiratory support interventions and care methods aimed at preventing hypothermia in preterm newborns reduce respiratory workload and help maintain more stable body temperature. Furthermore, the effects of non-invasive ventilation and nasal continuous positive airway pressure on body temperature in preterm infants requiring respiratory support have been examined, and it has been emphasized that the results need to be thoroughly evaluated in terms of thermoregulation.

In this context, our study aims to examine the relationship between body temperature and the characteristics, medical history, interventions performed within the first six hours, and follow-up findings of preterm newborns receiving respiratory support. By evaluating the relationships between variables in preterm infants receiving different types of respiratory support, a fundamental data model will be created that will contribute to optimizing practices aimed at maintaining thermoregulation. The results obtained may guide clinical practice by contributing to the development of appropriate thermoregulation management strategies in neonatal intensive care units, thereby reducing the risk of hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns born before 38 weeks of gestation and immediately admitted to the neonatal intensive care unit after birth
* who received respiratory support

Exclusion Criteria:

* Newborns who did not receive respiratory support immediately after birth despite being preterm at gestational age
* who have developmental health problems
* who have congenital health problems
* who were transferred from another healthcare facility after birth

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm newborns hospitalized in the Neonatal Intensive Care Unit at Acıbadem Healthcare Group Hospitals in Istanbul
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Change in body temperature | At birth and every hour for up to 6 hours after birth
  Body temperature measurement evaluated as axillary. Data for premature infants were collected hourly immediately after birth and for 6 hours following birth.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Kan Öntürk, Assoc. Prof., Principal Investigator — Acibadem University
Locations (1):
- Acıbadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Getaneh FB, Misganaw NM, Mihretie DB, Bitew ZW. Admission Hypothermia and Factors Associated with Mortality among Admitted Hypothermic Preterm Neonates in Neonatal Intensive Care Units of Public Hospitals of Addis Ababa, Ethiopia. Int J Pediatr. 2022 Oct 8;2022:8078628. doi: 10.1155/2022/8078628. eCollection 2022. PMID 36254265
- [Background] Feyisa GT, Marami SN, Dinagde DD, Degefe BD, Abebe ST, Kitil GW, Biratu AK. Comparative study of neonatal hypothermia and associated factors among neonates in rural and urban areas of the Shebadino Woreda, Sidama region, Southern Ethiopia: a community-based comparative cross-sectional study. BMC Public Health. 2024 Jul 20;24(1):1945. doi: 10.1186/s12889-024-19504-8. PMID 39033283
- [Background] Nyandiko WM, Kiptoon P, Lubuya FA. Neonatal hypothermia and adherence to World Health Organisation thermal care guidelines among newborns at Moi Teaching and Referral Hospital, Kenya. PLoS One. 2021 Mar 23;16(3):e0248838. doi: 10.1371/journal.pone.0248838. eCollection 2021. PMID 33755686
- [Background] Mohamed SOO, Ahmed SMI, Khidir RJY, Shaheen MTHA, Adam MHM, Ibrahim BAY, Elmahdi EOA, Farah ASM. Outcomes of neonatal hypothermia among very low birth weight infants: a Meta-analysis. Matern Health Neonatol Perinatol. 2021 Sep 15;7(1):14. doi: 10.1186/s40748-021-00134-6. PMID 34526138
- [Background] Demtse AG, Pfister RE, Nigussie AK, McClure EM, Ferede YG, Tazu Bonger Z, Mekasha A, Demisse AG, Gidi NW, Metaferia G, Worku B, Goldenberg RL, Muhe LM. Hypothermia in Preterm Newborns: Impact on Survival. Glob Pediatr Health. 2020 Sep 13;7:2333794X20957655. doi: 10.1177/2333794X20957655. eCollection 2020. PMID 32974416